CLINICAL TRIAL: NCT05904704
Title: Feasibility of Oxygen Enhanced MRI in Assessment of Malignant Brain Tumors
Brief Title: Oxygen-Enhanced MRI for Generating Hypoxia Maps in Patients With Intracranial Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ramon Barajas, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00025277; NCI-2023-01433 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025277 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (oxygen-enhanced MRI) (Experimental): Patients receive supplemental oxygen while undergoing standard of care MRI.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Oxygen Therapy

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Oxygen Therapy — Receive supplemental oxygen
  Other Names: supplemental oxygen therapy

SUMMARY:
This clinical trial evaluates the feasibility of performing oxygen-enhanced magnetic resonance imaging (MRI) to generate hypoxia maps in patients with intracranial tumors. Decreased levels of oxygen (hypoxia) is a hallmark of malignant brain tumors. Chronic hypoxia is a stimulator of blood vessel formation, which is required for tumor growth and spread. Hypoxia also limits the effectiveness of radiation and chemotherapy. MRI is an imaging technique that uses radiofrequency waves and a strong magnetic field rather than x-rays to provide detailed pictures of internal organs and tissues. The administration of inhaled oxygen allows for an increased MRI signal effect size. Oxygen-enhanced MRI may be a non-invasive method that can physiologically estimate tissue hypoxia. With a better understanding of the extent of tumor hypoxia, more effective and patient-specific therapies could be devised to halt malignant tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of generating hypoxia maps from oxygen MRI.

SECONDARY OBJECTIVES:

I. Evaluate the association between oxygen MRI hypoxia maps generated using T2* and T1 MRI sequences.

II. Evaluate the association between oxygen MRI hypoxia maps and progression free survival.

OUTLINE:

Patients receive supplemental oxygen while undergoing standard of care MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older) with a known or suspected intracranial tumor
* Able to provide informed written consent and/or acceptable surrogate capable of providing consent on the patient's behalf
* Legally authorized representative (LAR)-signed informed consent and assent obtained for those subjects identified as decisionally impaired
* Intracranial lesion known or suspected to be neoplastic greater than 10 mL as assessed by T2/fluid attenuated inversion recovery (FLAIR) magnetic resonance (MR) imaging
* Karnofsky performance score > 60 or Eastern Cooperative Oncology Group (ECOG) < 3 as assessed by referring clinician
* Planning to undergo or previously received therapeutic intervention for the intracranial tumor

Exclusion Criteria:

* Pregnant or breastfeeding
* Contraindication to supplemental oxygen administration, MRI, or intravenous gadolinium based contrast agents.

  * Claustrophobia
  * Weight greater than modality maximum capacity
  * Presence of metallic foreign body or implanted medical devices in body not documented as MRI safe according to the Oregon Health & Science University (OHSU) Department of Radiology guidelines (including but not limited to cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
  * Sickle cell disease
  * Unsure of pregnancy status as assessed by Department of Radiology and Advanced Imaging Research Center (AIRC) guidelines
  * Subjects for whom supplemental oxygen could be harmful such as people with potential for hypoventilation or chronic respiratory insufficiency (end-stage chronic obstructive pulmonary disease [COPD], obstructive sleep apnea [OSA] on continuous positive airway pressure [CPAP]/biphasic positive airway pressure [Bi-PAP], etc)
  * Subjects with a relative contraindication to supplemental oxygen administration will not be provided oxygen but may still participate in the study
* Presence of any other co-existing condition that, in the judgment of the principal investigator, might increase the risk to the subject (i.e., plans for hospice or end of life care)
* Poor peripheral intravenous access evaluated by patient history
* Presence of other serious systemic illnesses, including: uncontrolled infection, other uncontrolled malignancy, uncontrolled diabetes type II, or psychiatric/social situations which might impact the endpoint of the study or limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Generation of whole brain oxygen magnetic resonance imaging (MRI) data set | One hour of diagnostic imaging
  Evaluated to determine the feasibility of obtaining oxygen MRI hypoxia maps. Following completion of cohort enrollment, the generation of each hypoxia map will be independently scored as a dichotomous variable; successful or non-successful. The successful generation of a hypoxia map from either a T1 or T2* approach in 85% of the cohort of patients will need to be achieved for the imaging modality to be deemed feasible for the purposes of this study. Will provide the estimated proportion of success rate for each metric along with the corresponding 95% exact confidence interval.
Quantification of hypoxic tumor volume | One hour of diagnostic imaging
  Evaluated to determine the feasibility of obtaining oxygen MRI hypoxia maps.

SECONDARY OUTCOMES:
Correlation between T1 and T2* sequence hypoxia volume | One hour of diagnostic imaging
  Will determine the association between oxygen MRI hypoxia maps generated using T2* and T1 MRI sequences. Assessed using Pearson's correlation coefficient.
Progression free survival | Clinical follow up for up to 5 years
  Will perform Kaplan Meier analysis of progression free survival stratified by median T1 and T2* hypoxic volume to determine the association between oxygen MRI hypoxia maps and progression free survival. A Cox regression model will also be explored by treating hypoxic volume as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Barajas, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States